CLINICAL TRIAL: NCT06859476
Title: Study of Non-inferiority Between Manzanilla Sophia® and Meticel Ofteno® 0.5% for Providing a Relief Sensation to the Eyes
Brief Title: Evaluation of Manzanilla® and Meticel Ofteno® 0.5% for Providing a Relief Sensation to the Eyes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SOPHMAN-0824/IV
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Ophthalmological Agent Toxicity
Keywords: Matricaria Recutita

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manzanilla Sophia® (Experimental): Matricaria recutita 0.025%. One drop four times per day (QID), with a minimun interval of 3 hours between administrations, for 7 days.
  Interventions: Drug: Manzanilla Sophia®
- Meticel Ofteno® 0.5% (Active Comparator): Hydroxypropyl methylcellulose 0.5%. One drop QID, with a minimun interval of 3 hours between administrations, for 7 days.
  Interventions: Drug: Meticel Ofteno® 0.5%

INTERVENTIONS:
Drug: Manzanilla Sophia® — Ophthalmic solution. Laboratorios Sophia, S.A. de C.V., Zapopan, Jalisco, Mexico.
  Route of Administration: Ophthalmic.
  Arms: Manzanilla Sophia®
Drug: Meticel Ofteno® 0.5% — Ophthalmic solution. Laboratorios Sophia, S.A. de C.V., Zapopan, Jalisco, Mexico.
  Route of Administration: Ophthalmic.
  Arms: Meticel Ofteno® 0.5%

SUMMARY:
Demonstrate the non-inferiority of Manzanilla Sophia® compared to Meticel Ofteno® 0.5% in providing a sensation of eye relief, through the score of an analogous visual test for eye fatigue.

DETAILED DESCRIPTION:
Primary Objective:

Demonstrate the non-inferiority of Manzanilla Sophia® compared to Meticel Ofteno® 0.5% in providing a sensation of eye relief, through the score of an analogous visual test for eye fatigue.

Secondary Objectives:

Signs and Symptoms Evaluated:

* Compare Manzanilla Sophia® to Meticel Ofteno® 0.5% in the incidence of red eye.
* Compare Manzanilla Sophia® to Meticel Ofteno® 0.5% in the incidence of dry eye sensation.
* Compare Manzanilla Sophia® to Meticel Ofteno® 0.5% in the incidence of eye irritation.
* Compare Manzanilla Sophia® to Meticel Ofteno® 0.5% in the incidence of sensation of eye discharge (sleep).
* Compare Manzanilla Sophia® to Meticel Ofteno® 0.5% in the incidence of comfort with the application of the investigational product (IP).

Safety Assessment:

- Compare the incidence of adverse events (AEs) related to the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Ability to voluntarily provide signed informed consent.
* Able and willing to comply with the scheduled visits, treatment plan, and other study procedures.
* Be of legal age.
* Women of reproductive age who have not undergone bilateral tubal ligation or hysterectomy must ensure the continued use (initiated ≥ 30 days prior to signing the - - Informed Consent Form [ICF]) of a hormonal contraceptive method or intrauterine device (IUD) during the study period.
* A score of ≥ 3 on the analogous visual test for eye fatigue in at least 4 of the included questions.

Exclusion Criteria:

* Pregnant women, breastfeeding women, or those planning to become pregnant during the study period.
* Having participated in another clinical research study ≤ 30 days prior to the screening visit.
* Having previously participated in this study.
* Having only one functional eye.
* A history of current or past drug addiction or substance dependence within the last two years prior to signing the ICF.
* Current user of soft or hard contact lenses. They may be included if they suspend use during the study, and they must be lens-free for 15 days prior to inclusion.
* Known hypersensitivity to the components of the investigational products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2025-05-23 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
To demonstrate the non-inferiority of Manzanilla Sophia® compared to Meticel Ofteno® 0.5% in providing a sensation of eye relief, through the score of an analogous visual test for eye fatigue | Day 0 (Basal visit), Day 8 (Final visit)
  Score of the analogous visual test for eye fatigue. Based on other tools previously used for the assessment of eye fatigue, the visual analog test for eye fatigue used in this protocol is adapted and created. This test includes the following questions: "Have you had a headache?", "Have you had eye strain?", "Do you have gritty sensation in your eyes?", "Have your eyes been itchy?", "How would you describe your clarity of sight?", "Do you feel any discomfort when you fix your eyes?". Each of these questions will be answered according to a Likert scale of 1-5. The sum of the answers, the total score, will be measured in a scale from 6 to 30. A higher score is a a worse outcome for this variable.

SECONDARY OUTCOMES:
Comparison of Manzanilla Sophia® and Meticel Ofteno® 0.5% in the incidence of red eye | Day 0 (Basal visit), Day 8 (Final visit)
  Number of cases of red eye
Comparison of Manzanilla Sophia® and Meticel Ofteno® 0.5% in the incidence of dry eye sensation. | Day 0 (Basal visit), Day 8 (Final visit)
  Number of cases of dry eye sensation
Comparison of Manzanilla Sophia® and Meticel Ofteno® 0.5% in the incidence of eye irritation | Day 0 (Basal visit), Day 8 (Final visit)
  Number of cases of eye irritation sensation
Comparison of Manzanilla Sophia® and Meticel Ofteno® 0.5% in the incidence of sensation of eye discharge. | Day 0 (Basal visit), Day 8 (Final visit)
  Number of cases of sensation of eye discharge (sleep)
Comparison of Manzanilla Sophia® and Meticel Ofteno® 0.5% in the incidence of comfort with the application of the investigational product (IP). | Day 0 (Basal visit), Day 8 (Final visit)
  Number of cases of comfort after the application of the investigational product (IP)

OTHER OUTCOMES:
Comparison of the incidence of adverse events (AEs) related to the interventions between groups | Day 0 (Basal visit), Day 8 (Final visit)
  Number ofAEs related to the interventions

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad Clinica de Bioequivalencia (UNEBI), S de R.L de C.V., Guadalajara, Jalisco, Mexico